CLINICAL TRIAL: NCT06879366
Title: Evaluation of the Efficacy of Aloe-Vera el Versus Bezydamine Hydrochloride in the Treatment of Radiation Induced Oral Mucositis A Randamized Controlled Clinical Trial
Brief Title: Evaluation of the Efficacy of Aloe-Vera el Versus Bezydamine Hydrochloride in the Prevention of Radiation Induced Oral Mucositis A Randamized Controlled Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Amira Abdelwhab, lecturer of oral medicine, diagnosis and periodontology, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N-205-2023
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Cancer Patients Treated With Radiotherapy
MeSH Terms: interventions — Aloe vera gel; Benzydamine; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group: Aloe vera gel (Active Comparator)
  Interventions: Drug: Aloe vera gel
- control group: enzydamine gel (Active Comparator)
  Interventions: Drug: Benzydamine Hydrochloride 0.15% Oral gel

INTERVENTIONS:
Drug: Aloe vera gel — 10% aloe-vera gel will be prepared under well-controlled laboratory checks
  Arms: intervention group: Aloe vera gel
Drug: Benzydamine Hydrochloride 0.15% Oral gel — Benzydamine Hydrochloride 0.15% Oral gel
  Arms: control group: enzydamine gel

SUMMARY:
Background and Rationale Oral mucositis (OM) is one of the most debilitating toxic side effects of radiotherapy and chemotherapy. ]Radiation-induced OM occurs due to the generation of free radicals, which induce mitochondrial dysfunction resulting in increased oxidative stress, DNA damage and cell apoptosis. Epidermal growth factor (EGF) levels were decreased in patients with severe OM, and patients with lower levels of EGF prior to therapy may indicate increased risk of mucosal damage during RT

Objectives:

The purpose of this study is for Evaluation of the efficacy of aloe-vera gel versus standard treatment as a new option in the treatment of radiation-induced oral mucositis

Study population & Sample size :

40 patient proven to have Head and neck cancer , requiring radiotherapy.

Study Design:

RCT. The patients are randomized and divided into 2 groups , group A will use alovera gel , Group B will use benzylamide gel, EGF will be measured in saliva before and after 4 weeks treatment Methods Patient's visits will be at baseline, 2 weeks and 4 weeks. At follow up visits patients will be instructed to bring back the consumed container to check that they had totally consumed their previous supply before giving them the new one. Saliva collection to measure EGF by ELIZA

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients who are diagnosed with radiation-induced oral mucositis with any of its grades as scored by the world health organization (WHO) oral mucositis grading scale.

Exclusion Criteria:

* patients under the age of 18 ,patients receiving any previous treatment for oral mucositis during the last 2 weeks, allergy to aloe-vera, patients with chronic liver disease, infectious diseases (HIV, HBV,HCV,….), immune system dysfunction, haematological diseases and pregnancy or breast-feeding

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
1) Mucositis score | 0, 2 weeks , weeks, 6 weeks and 10 weeks
  1) Mucositis score which was recorded and graded as recommended by WHO . The grading criteria are as follows: grade 0 - no changes; grade I - soreness/(+)erythema; grade II - erythema (++), ulcer, can eat food(erythema with ulcers less than 1 cm2); grade III - ulcer(+++), (erythema with ulcers more than 1 cm2), requires liquid food; and grade IV - ulcer with haemorrhage and necrosis, alimentation not possible.
pain score | 0, 2,4,6, and 10 weeks
  2) Pain was recorded recommended by the Lindquist/Hickey scale 0 (none)- no pain; 1 (mild) - slight burning; 2 (moderate) - oral pain but able to eat; and 3 (severe) - severe pain and unable to eat.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt